CLINICAL TRIAL: NCT03297320
Title: Advance Care Planning at London Health Sciences Centre
Acronym: ACP@LHSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-16-299
Record Dates: First submitted 2017-09-26; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Advance Care Planning
Keywords: Advance Care Planning, End of life, CPR
MeSH Terms: conditions — Death

STUDY DESIGN:
Intervention Model Description: Healthcare teams in Internal Medicine at London Health Sciences Centre will be asked if they have any patients that need further goals of care discussions or ACP.
  A random selection of Internal Medicine patients will also be selected for further indepth conversations related to goals of care discussions or ACP
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team Referrals (Active Comparator): In-depth conversations about Goals of Care and ACP (the intervention) will be held for the patients referred to the research team by the three healthcare teams in Internal Medicine at London Health Sciences Centre (University Campus)
  Interventions: Other: In-depth conversation about Goals of Care and ACP
- Random selection (Active Comparator): A random selection of patients (not referred to the research team by the healthcare team) in Internal Medicine at London Health Sciences Centre (University Campus) will be selected to have in-depth conversations about Goals of Care and ACP (the intervention)
  Interventions: Other: In-depth conversation about Goals of Care and ACP

INTERVENTIONS:
Other: In-depth conversation about Goals of Care and ACP — In-depth conversation regarding Goals of Care and ACP by an experienced practitioner

SUMMARY:
All patients admitted to London Health Sciences Centre (LHSC) are asked to indicate their preferences for CPR (cardiopulmonary resuscitation) and other life-sustaining treatments that necessitate an Intensive Care Unit (ICU) admission.

Complex, high-risk patients at LHSC require multiple admissions to the hospital towards their end-of-life (EOL). Documentation of their resuscitation status should be a part of a broader dialogue with patients around their goals of care (GOC) and advance care planning (ACP), but rarely is this the case.

The innovation will involve the use of trained nurse facilitators to have meaningful conversations with patients and their families in an effective way that bridges the gap between resuscitation status, GOC discussions and ACP across the continuum of care.

DETAILED DESCRIPTION:
1. On admission, the usual LHSC process will be followed whereby the patient's wishes for resuscitation are documented on the resuscitation record in the patient's chart. This constitutes the "original" resuscitation status.
2. After referral or screening and written consent, the RA will conduct semi-structured, face-to-face interviews with the patient and or SDM as appropriate. If the RA has concern about a discordance, he/she will then provide verbal feedback to the health-care team (Attending Physician or the Senior Medical Resident (SMR)) immediately and request them to communicate with the patient/SDM again. A case of discordance shall be recorded ONLY if the health-care team (Attending Physician or Senior Medical Resident) confirms that a change in resuscitation status is needed. The output of this intervention will be the "revised" resuscitation status. This "standardized" process for determining this outcome has worked well in our pilot study. Any disagreements between RA and SMR on patient/SDM preferences will be reported to Team#1 Attending and recorded. It will be up to the team to reconcile the "revised" resuscitation preferences on official records (Resuscitation status can only be filled in only by an MD as per hospital policy).

4. Advanced Clinical Notes: These will be typed by the RA and a note be made of the "revised" resuscitation preferences along with GOC and ACP discussions.

5. A pilot study related to this work started in August 2016 and has allowed the research team to evaluate barriers and facilitators of conducting this intervention on Internal Medicine patients.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to internal medicine teams at or after hospitalization day 2 with:

1. Age ≥55 years with ≥1 diagnoses: Chronic lung disease, Coronary artery disease, Congestive heart failure, Cirrhosis, Renal failure, Diabetes, Peripheral vascular disease, Cancer, Dementia (inability with ADLs) or
2. If none of these criteria were met, any patient whose death within the next 1 year would not surprise health-care team members.

Exclusion Criteria:

1. Lack of written consent
2. Patients who do not speak English; hard of hearing
3. Expected to die or be discharged ≤ 24 hours
4. Referral to or having an established palliative care plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Discordance | 2 years
  Discordance between patients' prior expressed preferences and those documented in their healthcare record

SECONDARY OUTCOMES:
Risk factors associated with discordance | 2 years
  Evaluate predisposing factors for the discordance

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Taneja, FRCPC, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No